CLINICAL TRIAL: NCT00090428
Title: Diet and Behavior in Young Children With Autism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, susan hyman, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U54MH066397 (NIH); U54MH066397 (NIH); DDTR BD-DD
Record Dates: First submitted 2004-08-26; First posted 2004-08-27 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Autism; Autistic Disorder
Keywords: Autism; Applied Behavioral Analysis; Gluten; Casein
MeSH Terms: conditions — Autistic Disorder | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will follow a gluten-free and casein-free diet for 18 weeks. The compliance with the diet was monitored with 24 hour dietary recall and nutritional sufficiency with diet diary analysis.
  Interventions: Behavioral: Gluten- and casein-free diet
- 2 (Active Comparator): After established on a gluten free and casein free diet for at least 6 weeks, participants received double blind, placebo controlled challenges containing gluten, casein, gluten+casein, or placebo in a random order. Data was collected on behavioral and physiologic responses relative to the challenges. Children remained on the gluten free and casein free diet throughout this period.
  Interventions: Behavioral: Placebo controlled diet

INTERVENTIONS:
Behavioral: Gluten- and casein-free diet — Participants will follow a gluten-free and casein-free diet for 18 weeks. All children received individual EIBI interventions to decrease the confound of different types of therapies.
  Arms: 1
Behavioral: Placebo controlled diet — Participants will follow a gluten-free and casein-free diet for 18 weeks. They will receive double blind placebo controlled challenge snacks that contain gluten, casein, gluten+casein or placebo with measurement of response. They remain on the gluten free and casein free diet for the entire study period.
  Arms: 2

SUMMARY:
This study will determine whether a gluten- and casein-free diet has specific benefits for children with autism.

DETAILED DESCRIPTION:
Autism is a serious brain disorder that affects brain development and often causes social and educational problems. Prior studies suggested that a gluten- and casein-free diet may have a therapeutic effect on the behavior of children with autism. This study will examine the effects of such a diet on the behavior of children with autism who meet research diagnostic criteria, are monitored in adherence to the diet, and receive similar intense behavioral therapy.

Children in this study will be following a gluten free and casein free diet for 18 weeks. All subjects will have 6 weeks of baseline followed by 12 weeks of randomized, double-blind, placebo-controlled, challenge snacks with careful behavioral observation and evaluation. They also will be receiving uniform educational and behavioral services through their provider. Standard autism evaluation methods, weekly diet and sleep diaries and scheduled laboratory tests will be used to assess subjects. An end of study, follow-up assessment will be completed at 30 weeks after the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Autism spectrum disorder or pervasive developmental disorder, ADI-R and ADOS positive.
* Participation in applied behavioral analysis classes for at least 4 months, with at least 10 hours per week of service, and at least 1 hour of service in the home
* A score higher than 30 on the Mullen Early Learning scale
* Ability to maintain a gluten- and casein-free diet during the study
* In order to maintain study integrity, and due to frequent child assessments, enrollment is limited to a select population within the Rochester area

Ages: 30 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2004-01; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of the gluten free casein free diet | Measured at Weeks 6,18 and 30
  Behavioral data: activity, sleep, behaviors related to the autism; Medical data: stool pattern, nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hyman, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States